CLINICAL TRIAL: NCT03292575
Title: Prevention of Cardio-embolic Stroke Using Anti-vitamin K and Direct Oral Anticoagulants. A Model of Action in Burgundy.
Brief Title: Study of the Follow-up of Stroke Treated With Anticoagulants
Acronym: AOD
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: Giroud 2016
Record Dates: First submitted 2017-09-21; First posted 2017-09-25 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Anticoagulants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stroke related to CAAF
  Interventions: Drug: Anticoagulants

INTERVENTIONS:
Drug: Anticoagulants

SUMMARY:
Stroke is a major public health problem as it is very frequent (140,000 cases/year in France), and very serious (leading cause of death, 2nd leading cause of dementia, 3rd leading cause of handicap). Ischemic cardio-embolic stroke accounts for around 25% of ischemic strokes, and ischemic cardio-embolic stroke in a context of cardiac arrhythmia due to atrial fibrillation (CAAF) is the leading non-atheromatous cause. The aim of this study is to optimise the secondary prevention of CAAF-related stroke identified at the University Hospital of Dijon Burgundy in the framework of the recommendations of the '2010-2014 stroke plan' and the Compulsory Consultation at the 6th month (Directive DGOS//2015/262 of the 3rd August 2015)

ELIGIBILITY:
Inclusion Criteria:

* patients managed for stroke at the stroke unit of Dijon University Hospital for CAAF-related cardio-embolic stroke

Exclusion Criteria:

* NA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patient with stroke resulting from occlusion of a cerebral artery (cerebral infarction) with a clot detached from the heart that exhibits an arrhythmia by Auricular Fibrillation or the occurrence of intracerebral hemorrhage
Sampling Method: Probability Sample
Enrollment: 441 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
rate of stroke recurrences | 12 months after inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France